CLINICAL TRIAL: NCT06521580
Title: What Are the Clinical and Radiological Outcomes of Open Reduction and Internal Fixation in Adult Patients With Osteopetrosis Weight-bearing Bone Fractures
Brief Title: Outcomes of Patients With Osteopetrosis Weight-bearing Bone Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, Dr., Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-375-2023
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Osteopetrosis
MeSH Terms: conditions — Osteopetrosis | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open reduction and internal fixation (Experimental): Open reduction and internal fixation (ORIF) is a common surgical technique used to treat fractures by realigning and stabilizing the broken bones with hardware such as plates, screws, or rods. In the context of osteopetrosis, ORIF can be particularly challenging due to the sclerotic nature of the bone, which makes drilling and hardware placement difficult, and the poor vascularity, which can impede healing and increase the risk of complications such as nonunion or infection.
  Interventions: Procedure: Open reduction and internal fixation

INTERVENTIONS:
Procedure: Open reduction and internal fixation — Open reduction and internal fixation of those with osteopetrosis and weight bearing fractures

SUMMARY:
Osteopetrosis is a rare genetic disorder characterized by the abnormal hardening and density of bones, leading to increased brittleness and susceptibility to fractures. This condition presents significant challenges in fracture management due to the altered bone architecture and compromised healing capacity. Open reduction and internal fixation (ORIF) is a common surgical technique employed to stabilize fractures, but its efficacy and outcomes in patients with osteopetrosis are not well-documented. This study aims to evaluate the clinical and radiological outcomes of ORIF in adult patients with weight-bearing bone fractures due to osteopetrosis, providing insights into the effectiveness and potential complications of this treatment approach.

DETAILED DESCRIPTION:
Osteopetrosis, also known as marble bone disease, is a rare genetic disorder that leads to the abnormal hardening and densification of bones due to defective osteoclast-mediated bone resorption. This imbalance results in bones that are abnormally dense yet fragile and prone to fractures. Osteopetrosis is typically categorized into three major types based on severity and inheritance patterns: autosomal recessive infantile osteopetrosis, autosomal recessive intermediate osteopetrosis, and autosomal dominant adult osteopetrosis.

In adult patients, osteopetrosis often presents with a range of clinical manifestations including bone pain, frequent fractures, cranial nerve compression, and hematological abnormalities due to bone marrow space reduction. Weight-bearing bones such as the femur, tibia, and pelvis are particularly susceptible to fractures due to the mechanical stress they endure. These fractures pose significant clinical challenges because the dense bone structure complicates surgical intervention and delays healing.

Open reduction and internal fixation (ORIF) is a common surgical technique used to treat fractures by realigning and stabilizing the broken bones with hardware such as plates, screws, or rods. In the context of osteopetrosis, ORIF can be particularly challenging due to the sclerotic nature of the bone, which makes drilling and hardware placement difficult, and the poor vascularity, which can impede healing and increase the risk of complications such as nonunion or infection.

Despite these challenges, ORIF remains a critical option for managing fractures in osteopetrosis patients. Understanding the clinical and radiological outcomes of this intervention can help optimize treatment protocols and improve patient care. This case series aims to evaluate the outcomes of ORIF in adult patients with osteopetrosis-induced weight-bearing bone fractures. By examining factors such as fracture healing, functional recovery, and complication rates, this study seeks to provide valuable insights into the effectiveness and potential risks associated with ORIF in this unique patient population.

ELIGIBILITY:
Inclusion Criteria:

All patients with adult osteopetrosis above 18 years of age

Exclusion Criteria:

Non-weight-bearing fractures Non-osteopetrosis patients Pediatric patients Previous fracture surgery Concurrent bone conditions Inability to follow up Infection at fracture site Severe comorbidities Pregnancy Non-surgical treatment preference

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Bone union | 6 months
  We follow up the patients for bone union through radiological examination

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy-Cairo University- Faculty of Medicine, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
unless upon reasonable request